CLINICAL TRIAL: NCT05226039
Title: The Effects of a Single Bout of Aerobic Exercise on Cognition: The Moderating Role of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: North American Society for the Psychology of Sport and Physical Activity (Unknown)
Responsible Party: Principal Investigator, Jarod Vance, Principal Investigator, University of North Carolina, Greensboro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FY22-134
Record Dates: First submitted 2021-10-04; First posted 2022-02-07 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cognitive Performance

STUDY DESIGN:
Intervention Model Description: Following the first visit, participants will be randomly counterbalanced to one of the two conditions first (exercise, or control condition). Following completion of the first condition, the third visit will be completion of the other condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young adult group (Other): One group will consist of 20 to 30 year olds. Participants will complete all three visits that include both the treatment (exercise visit) and the control (rest) visits. The treatment visit will consist of 20 minutes of moderate intensity aerobic exercise on a stationary bike.
  Interventions: Behavioral: Moderate intensity acute exercise bout
- Older adult group (Other): The other group will consist of 60 to 70 year olds. Participants will complete all three visits that include both the treatment (exercise visit) and the control (rest) visits. The treatment visit will consist of 20 minutes of moderate intensity aerobic exercise on a stationary bike.
  Interventions: Behavioral: Moderate intensity acute exercise bout

INTERVENTIONS:
Behavioral: Moderate intensity acute exercise bout — The treatment/intervention will consist of 20 minutes of moderate intensity aerobic exercise on a stationary bike. Intensity will be prescribed based off of heart rate reserve.

SUMMARY:
The current clinical study will have two groups of participants (young adults ages 20 - 30, and older adults ages 60 - 70) take part in three visits to the lab. On the first visit participants will fill out questionnaires assessing demographics and physical activity level. On the 2nd and 3rd visits participants will be engage in both a moderate intensity bout of aerobic exercise for 20 minutes, and 20 minutes of resting on a stationary bike watching an educational video. These two visits will be counterbalanced across age groups. Following both the exercise bout and the resting control condition participants will complete cognitive tasks assessing episodic memory and executive functioning. The first hypothesis is that older adults who are more physically active (assessed via questionnaire) will have significantly greater cognitive abilities compared to those who are less active or sedentary. The second hypothesis is that following a single bout of moderate intensity aerobic exercise, older adults will have a greater magnitude of change in their short-term memory, and long-term memory performance compared to younger adults.

DETAILED DESCRIPTION:
Participants who express interest in the study will be contacted by telephone. During this phone call, the primary investigator will assess the inclusion/exclusion criteria (i.e., investigators will ask their age, if participants are willing to stay inactive during the required times, refrain from caffeine and food intake within an hour of every visit). Eligible participants will be scheduled for their 1st visit. On the first day of participation in the study, participants will read and sign the informed consent, complete questionnaires, and (to further assess their eligibility for both parts of the study) participants will perform the Montreal Cognitive Assessment, fill out a physical activity questionnaire, and complete a health history form (American College of Sports Medicine). On visit 1 participants will also complete cognitive tasks measuring memory and executive functioning. Investigators will assess resting heart rate by having participants put on a heart rate monitor to record R-R intervals (to assess heart rate variability) at rest for 5 minutes. If participants meet the eligibility requirements assessed on visit 1 (> 90 mins of physical activity/week) participants will qualify and be scheduled for visits 2 and 3.

During visits 2 and 3, participants will put on a heart rate monitor so that investigators can record their heart rate during the two conditions. Participants will then perform one of two conditions in a counterbalanced order. Participants will either rest for 25 minutes while watching an educational video, do the memory task, complete tasks measuring executive functioning (Stroop color word task, spatial working memory task), and do the recall task; or exercise for 25 min, do the memory task, complete the executive functioning tasks and do the recall task. The memory task is the Auditory Verbal Learning Test (AVLT) which consists of hearing and recalling a list of 15 words (List A) 5 times, hearing and recalling a different list of 15 words (List B), and then recalling List A. Participants will be audio recorded during the memory task to ensure that accurate scoring can be completed. The executive functioning tasks (Stroop, Spatial working memory task) will involve participants responding to stimuli on a computer via a keyboard. The Stroop task requires participants to respond to the color of stimuli that come up on the screen and the Spatial working memory task requires participants to remember the position of varying numbers of dots. The recall task involves participants recalling List A and then being asked to identify from a list of words those that came from List A or List B (recognition). The exercise consists of 5-min of warm-up followed by 20 min of moderate intensity exercise (55-65% heart rate reserve at 60-80 revolutions per minute). All exercise and rest periods will be on a cycle ergometer. During all memory tasks, there will be audio-taping. Subjects will be scheduled with a minimum of 48 hours between Day 1 and Day 2 and between Day 2 and Day 3.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 30 years old for young adult group
* 60 to 70 years old for older adult group
* Cognitive normal (assessed via Montreal Cognitive Assessment on visit 1)

Exclusion Criteria:

* Do not have any contraindications to exercise (assessed via American College of Sport Medicine Health screening form)
* No current musculoskeletal injuries

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Episodic memory - Rey Auditory Verbal Learning Task Visit 1 | Approximately 20 minutes into visit 1.
  The Rey Auditory Verbal Learning task (RAVLT) will assess single-item episodic memory. The number of words correctly recalled on 8 trials will be measured.
Episodic memory - Rey Auditory Verbal Learning Task Visit 2 | immediately following exercise or control (witnin 5 minutes)
  The Rey Auditory Verbal Learning task (RAVLT) will assess single-item episodic memory. The number of words correctly recalled on 8 trials will be measured.
Episodic memory - Rey Auditory Verbal Learning Task Visit 3 | immediately following exercise or control (within 5 minutes)
  The Rey Auditory Verbal Learning task (RAVLT) will assess single-item episodic memory. The number of words correctly recalled on 8 trials will be measured.
Episodic memory - Associative memory task Visit 1 | Approximately 45 minutes into visiti 1.
  Participants will hear pairs of words read to them over an audio recording. Following this they will be asked to name the second word in each pair during recall. The number of words correctly recalled on 3 trials will be measured.

SECONDARY OUTCOMES:
Executive functioning - Stroop reaction time Visit 1 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Reaction time will be assessed.
Executive functioning - Stroop reaction time Visit 2 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Reaction time will be assessed.
Executive functioning - Stroop reaction time Visit 3 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Reaction time will be assessed.
Executive functioning - Stroop accuracy Visit 1 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Accuracy on the task will be assessed.
Executive functioning - Stroop accuracy Visit 2 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Accuracy on the task will be assessed.
Executive functioning - Stroop accuracy Visit 3 | Executive functioning will be measured 7 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Stroop Color Word task. Accuracy on the task will be assessed.
Executive functioning - Spatial working memory reaction time Visit 1 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Reaction time on this task will be measured.
Executive functioning - Spatial working memory reaction time Visit 2 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Reaction time on this task will be measured.
Executive functioning - Spatial working memory reaction time Visit 3 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Reaction time on this task will be measured.
Executive functioning - Spatial working memory accuracy Visit 1 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Accuracy on this task will be measured.
Executive functioning - Spatial working memory accuracy Visit 2 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Accuracy on this task will be measured.
Executive functioning - Spatial working memory accuracy Visit 3 | Executive functioning will be measured 12 minutes after completion of the exercise or control conditions.
  Executive functioning will be assessed using a Spatial Working memory task. Accuracy on this task will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
The current study is Jarod Vances' Dissertation project. A plan has not been created to share the data at this time due to the nature of the study having a very specific scope to be assessed.